CLINICAL TRIAL: NCT02898298
Title: Positive Emotion Regulation Training in Children, Adolescents and Young Adults With and Without Developmental Disorder
Acronym: ERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Andrea Samson, Senior Researcher, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-242
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Experimental): Immediate group receives the Positive Emotion Regulation training immediately.
  Interventions: Behavioral: Positive Emotion Regulation Training
- Waitlist control group (Active Comparator): Waitlist control group receives the Positive Emotion Regulation training 4 weeks later.
  Interventions: Behavioral: Positive Emotion Regulation Training

INTERVENTIONS:
Behavioral: Positive Emotion Regulation Training — Participants will receive a 3-session psycho-educative training on emotion regulation.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel positive emotion regulation intervention that aims to increase positive emotions and improve emotion regulation skills in children, adolescents and young adults. The study focuses on individuals with a developmental disorder such as Autism Spectrum Disorder and other Learning or Developmental Disabilities in comparison to typically developing (TD) controls. Participants will complete a psycho-educative training to learn about positive emotions and how to increase them in their daily lives. Participants are expected to benefit from the training, which will be evident in a change in emotion experience, emotion regulation strategy use, and well-being. Emotion regulation efficacy will be related to symptom severity (autistic symptoms), alexithymia and problematic behaviors.

DETAILED DESCRIPTION:
This study aims at testing the efficacy of a 3-session psycho-educative training on emotion regulation and wellbeing in children and adolescents with or without developmental disorders with a waitlist control group design. Specifically, we are interested to improve different aspects of emotions, such as emotion experience, regulation strategy use, and beliefs on the malleability of emotions. Given that most of the past and actual interventions focus on negative emotions, our training will allow participants to learn more about positive emotions, how they can increase them, and how they can benefit from them.

Individuals with a developmental disorder including Autism Spectrum Disorder (ASD) will be recruited via flyers in specialized institutions and schools. Individuals with typical development (TD) will be recruited via flyers in schools, universities, libraries, and in other public places. Participants will be randomly assigned to the training or waiting list group (control). Randomization will be stratified for the two populations (i.e. with and without a developmental disorder) and for age. Participants and one of their parents (if <18 years) will be asked to fill in questionnaires on emotion experience, emotion regulation, beliefs about the malleability of emotions, well-being, problematic behaviors, alexithymia, and ASD symptom severity at four time points. Some questionnaires will only be completed by parents. Participants will be asked to answer additional questions on their emotional experience and emotion regulation and to provide examples of their own emotional experience and emotion regulation during and after each of the training sessions.

Participants are expected to benefit from the intervention, which should become evident in the changes of the primary outcome measures (emotion experience, emotion regulation, beliefs about the malleability of emotions, well-being) and the secondary outcome measures (problematic behaviors, alexithymia, and ASD symptom severity) post-intervention and at 8-weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 10-35 years old, presenting or not a developmental disorder (e.g., autism).

Exclusion Criteria:

* Participants who are not able to understand the training instructions.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Scale | Week 1, Week 5, Week 9, Week 13 or 17
  Change in emotion experience. Week 13 for immediate group, Week 17 for waitlist group.
Change in Emotion Regulation Questionnaire | Week 1, Week 5, Week 9, Week 13 or 17
  Change in emotion regulation strategy use. Week 13 for immediate group, Week 17 for waitlist group.
Change in Satisfaction with Life Scale | Week 1, Week 5, Week 9, Week 13 or 17
  Change in well-being. Week 13 for immediate group, Week 17 for waitlist group.
Change in Subjective Happiness Scale | Week 1, Week 5, Week 9, Week 13 or 17
  Change in well-being. Week 13 for immediate group, Week 17 for waitlist group.

SECONDARY OUTCOMES:
Change in Toronto Alexithymia Scale | Week 1, Week 5, Week 9, Week 13 or 17
  Change in alexithymia scores. Week 13 for immediate group, Week 17 for waitlist group.
Change in Strength and Difficulties Questionnaire | Week 1, Week 5, Week 9, Week 13 or 17
  Change in problematic behavior. Week 13 for immediate group, Week 17 for waitlist group.
Change in Autism Spectrum Quotient | Week 1, Week 5, Week 9, Week 13 or 17
  Change in autism symptom severity. Week 13 for immediate group, Week 17 for waitlist group.

OTHER OUTCOMES:
Participants' experience and satisfaction with training (satisfaction questionnaire) | Week 13 or 17
  Week 13 for immediate group, Week 17 for waitlist group.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Samson, Dr, Principal Investigator — University of Geneva; David Sander, Prof, Study Chair — University of Geneva
Locations (1):
- Swiss Center for Affective Sciences (Campus Biotech, University of Geneva), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross JJ. Antecedent- and response-focused emotion regulation: divergent consequences for experience, expression, and physiology. J Pers Soc Psychol. 1998 Jan;74(1):224-37. doi: 10.1037//0022-3514.74.1.224. PMID 9457784
- [Background] Gross JJ (2014). Emotion regulation: Conceptual and empirical foundations. In J.J. Gross (Ed.), Handbook of emotion regulation (2nd ed.) (pp. 3-20). New York, NY: Guilford.
- [Background] Gross, JJ, Jazaieri, H. Emotion, emotion regulation, and psychopathology an affective science perspective. Clinical Psychological Science 2(4): 387-401, 2014.
- [Background] Mazefsky CA, Pelphrey KA, Dahl RE. The Need for a Broader Approach to Emotion Regulation Research in Autism. Child Dev Perspect. 2012 Mar 1;6(1):92-97. doi: 10.1111/j.1750-8606.2011.00229.x. Epub 2012 Jan 12. PMID 22639681
- [Background] Mazefsky CA, Herrington J, Siegel M, Scarpa A, Maddox BB, Scahill L, White SW. The role of emotion regulation in autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2013 Jul;52(7):679-88. doi: 10.1016/j.jaac.2013.05.006. Epub 2013 Jun 3. PMID 23800481
- [Background] Quoidbach J, Mikolajczak M, Gross JJ. Positive interventions: An emotion regulation perspective. Psychol Bull. 2015 May;141(3):655-93. doi: 10.1037/a0038648. Epub 2015 Jan 26. PMID 25621978
- [Background] Riediger M, Klipker, K. (2014). Emotion regulation in adolescence. In Handbook of emotion regulation (pp. 187-202). Guilford Press.
- [Background] Samson AC, Huber O, Gross JJ. Emotion regulation in Asperger's syndrome and high-functioning autism. Emotion. 2012 Aug;12(4):659-65. doi: 10.1037/a0027975. Epub 2012 May 28. PMID 22642342
- [Background] Samson AC, Huber O, Ruch W. Seven decades after Hans Asperger's observations: A comprehensive study of humor in individuals with Autism Spectrum Disorders. Humor, 26(3): 441-460, 2013.
- [Background] Samson AC, Hardan AY, Lee IA, Phillips JM, Gross JJ. Maladaptive Behavior in Autism Spectrum Disorder: The Role of Emotion Experience and Emotion Regulation. J Autism Dev Disord. 2015 Nov;45(11):3424-32. doi: 10.1007/s10803-015-2388-7. PMID 25711546
- [Background] Samson AC, Hardan AY, Podell RW, Phillips JM, Gross JJ. Emotion regulation in children and adolescents with autism spectrum disorder. Autism Res. 2015 Feb;8(1):9-18. doi: 10.1002/aur.1387. Epub 2014 May 23. PMID 24863869
- [Background] Samson AC, Phillips JM, Parker KJ, Shah S, Gross JJ, Hardan AY. Emotion dysregulation and the core features of autism spectrum disorder. J Autism Dev Disord. 2014 Jul;44(7):1766-72. doi: 10.1007/s10803-013-2022-5. PMID 24362795
- [Background] Weytens F, Luminet O, Verhofstadt LL, Mikolajczak M. An integrative theory-driven positive emotion regulation intervention. PLoS One. 2014 Apr 23;9(4):e95677. doi: 10.1371/journal.pone.0095677. eCollection 2014. PMID 24759870
- [Derived] Zaharia A, Noir-Kahlo K, Bressoud N, Sander D, Dukes D, Samson AC. Proof of Concept: A Brief Psycho-Educational Training Program to Increase the Use of Positive Emotion Regulation Strategies in Individuals With Autism Spectrum Disorder. Front Psychol. 2021 Nov 1;12:705937. doi: 10.3389/fpsyg.2021.705937. eCollection 2021. PMID 34790142